CLINICAL TRIAL: NCT06339359
Title: A Pilot Study to Develop a Behavior-based Screening Protocol for Early Diagnosis of Autism Spectrum Disorders
Status: Recruiting | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2024-02-014
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: ASD
MeSH Terms: interventions — Kinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exmainations including clinical measurement, kinetic and kinematic measurmetns. Behavioral assessments — Collection of clinical data including K-Bayley Scales of Infant and Toddler Development Third Edition (K-BSID-Ⅲ), , Beery-Buktenica Visual-Motor Integration, Sixth Edition (VMI-6) and clinical measurement. motor analysis and eye tracking

SUMMARY:
This study aims to collect basic data to develop a tool for early screening of autism spectrum disorder (ASD) in children and adolescents through eye tracking and motion analysis.

DETAILED DESCRIPTION:
This study aims to collect basic data to develop a tool for early screening of autism spectrum disorder (ASD) in children and adolescents through eye tracking and motion analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents under the age of 19 at the time of registration
* A person whose legal representative voluntarily decides to participate and agrees in writing to comply with the precautions after receiving a detailed explanation of this study and fully understanding it

Exclusion Criteria:

* Those with abnormalities in hearing and vision
* Those who are likely to have difficulty participating in the study according to the judgment of the clinical investigator
* If the visits set out in this research plan are not followed or the patient's guardian does not cooperate due to low understanding of the patient.

Max Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
K-BSID-Ⅲ | Between March 2024 and March 2025
  Measurement of K-BSID-Ⅲ is a developmental test administered to infants from 16 days old to 42 months old, and consists of 16 subtests measuring a total of 5 development areas (cognitive, language, motor, social-emotional, and adaptive behavior).
ADI-R | Between March 2024 and March 2025
  Measurement of ADI-R is a test conducted to screen autism spectrum disorder from other developmental disabilities in children with a mental age of 2 years or older, and is conducted through a structured interview with the primary caregiver.
M-CHAT | Between March 2024 and March 2025
  Measurement of M-CHAT is a tool to screen the risk level of autism spectrum disorder in children aged 16 to 30 months and is evaluated based on the primary caregiver's report.
ADOS-2 | Between March 2024 and March 2025
  Measurement of ADOS-2 is a standardized assessment tool that evaluates social interaction and stereotyped and repetitive behavior in people suspected of having autism spectrum disorder.
K-WPPSI-Ⅳ | Between March 2024 and March 2025
  Measurement of K-WPPSI-Ⅳ is an intelligence test to evaluate cognitive function in children aged 2 years and 6 months to 7 years and 7 months.
K-CARS-2 | Between March 2024 and March 2025
  Measurement of K-CARS-2 is an one of the most widely used tools for the purpose of distinguishing autism from other developmental disabilities and the degree of autism.
CBCL | Between March 2024 and March 2025
  Measurement of CBCL is a useful clinical tool used in many countries around the world to evaluate social adaptation and emotional behavior problems in children and adolescents.
SCQ | Between March 2024 and March 2025
  Measurement of SCQ is a tool to screen symptoms related to autism spectrum disorder through parent report.
GMFM | Between March 2024 and March 2025
  Measurement of GMFM is a standardized observational evaluation tool with validity that measures changes in gross motor function over time in children with cerebral palsy.
HFT | Between March 2024 and March 2025
  Measurement of HFT is a tool to evaluate the degree of development of hand function according to age, forward arm reaching, various grasping abilities, coordination ability between both hands, and object handling ability.
BOT-2 | Between March 2024 and March 2025
  Measurement of BOT-2 is a testing tool used for movement training evaluation and development.
VMI-6 | Between March 2024 and March 2025
  Measurement of VMI-6 is a test that validly measures the visual-motor integration ability, visual perception ability, and motor coordination ability of various age groups from infants to adults.
SP | Between March 2024 and March 2025
  Measurement of SP is a standardized tool for assessing children's sensory processing patterns in the context of everyday life, providing unique information about how sensory processing supports or hinders participation.
Eye Tracking | Between March 2024 and March 2025
  While the subject watches the video material being played, gaze and behavioral data are recorded.
Motion Analysis | Between March 2024 and March 2025
  Measurement of Motion analysis is an evaluation process of the research subject is filmed while administering ADOS and RBS-EC.

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea